CLINICAL TRIAL: NCT03991520
Title: Pilot Study of the IL-1 Antagonist Anakinra for the Treatment of Endometriosis Related Symptoms
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sanjay Agarwal, Professor and Director of Fertility Services, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 182006
Record Dates: First submitted 2019-05-27; First posted 2019-06-19 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Endometriosis; Anakinra; Markers of Inflammation
MeSH Terms: conditions — Endometriosis | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment with Anakinra (Experimental): 10 subjects will be enrolled in this group. Initial treatment will consist of 100mg/day Anakinra, which is the standard, FDA approved dose for the treatment of rheumatoid arthritis. The randomized treatment will be self-administered by the subject each evening by subcutaneous injection from within 24 hours of the onset of menses until within 24 hours of last menstrual day.
  Interventions: Drug: Anakinra 100Mg/0.67Ml Inj Syringe
- Standard Comparison (Placebo Comparator): 10 subjects will be enrolled in this group. This group will be given placebo injections as their initial treatment. The placebo is comparable to the anakinra formulation without the active medication - a solution (pH 6.5) containing anhydrous citric acid (1.29 mg), disodium EDTA (0.12 mg), polysorbate 80 (0.70 mg), and sodium chloride (5.48 mg) in water for injection. These individuals will self-administer the placebo each evening by subcutaneous injection from within 24 hours of the onset of menses until within 24 hours of last menstrual day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anakinra 100Mg/0.67Ml Inj Syringe — The study drug is100mg/day Anakinra, which is the standard, FDA approved dose for the treatment of rheumatoid arthritis. The randomized treatment will be self-administered by the subject each evening by subcutaneous injection.
  Other Names: Kineret
  Arms: Active Treatment with Anakinra
Drug: Placebo — The placebo is comparable to the anakinra formulation without the active medication - a solution (pH 6.5) containing anhydrous citric acid (1.29 mg), disodium EDTA (0.12 mg), polysorbate 80 (0.70 mg), and sodium chloride (5.48 mg) in water for injection
  Arms: Standard Comparison

SUMMARY:
All current FDA approved medications to treat endometriosis pain including danazol, GnRH agonists (Lupron, Zoladex and Synarel), GnRH antagonist (elagolix) and depo-provera prevent or contradict pregnancy. Therefore women suffering from endometriosis and trying to conceive have no medical options apart from pain meds. The purpose of this pilot study is to determine whether the anti-inflammatory, IL-1 inhibitor (anakinra) reduces pelvic pain due to endometriosis without altering menstrual cycles, which is an indicator of ovulatory function. Anakinra is an FDA approved injectable medication for the treatment of rheumatoid arthritis that is pregnancy category B.

DETAILED DESCRIPTION:
Endometriosis is a chronic inflammatory disease1 that affects 5 -10% of reproductive aged women1,2. It is characterized by the presence of uterine endometrium outside the uterus. The condition causes health distress through pelvic pain and decreased QOL. Current therapies to temporarily control symptoms include surgery as well as medical options that prevent pregnancy and have significant side-effects.3,4 The most common symptoms with endometriosis include dysmenorrhea, dyspareunia and NMPP. Ultimately these lead to a decrease in QOL. All current medical therapies to treat endometriosis pain prevent or contradict pregnancy.

Inflammation is a well-established central figure in the pathophysiology of endometriosis(1). Increasingly, data is suggesting that IL-1 is a mediator of inflammation in endometriosis (2, 3). In addition, there are data that single nucleotide polymorphisms at the IL-1A gene locus are associated with endometriosis risk (4). Hence, it is rational to assess anakinra, an IL-1 antagonist, in the control of symptoms and inflammation due to endometriosis. Therefore, we propose this pilot study testing an FDA approved medication (anakinra) to reduce IL-1 and on dysmenorrhea due to endometriosis without stopping periods (a sign of ovulation).

Anakinra is a self-administered subcutaneous injectable medication that is FDA approved for the treatment of rheumatoid arthritis. As an IL-1 antagonist, it works by decreasing inflammation and is administered daily by the patient. Because Anakinra interferes with the immune system functioning, the major concern with the use of Anakinra is reduced resistance to infection. Others include injection site reactions such as redness, itching, rash, and pain. Bruising or bleeding also can occur, but it is rare. These effects usually stop after one - two weeks. Headaches and low white blood cell counts can also occur, but these are very rare. Anakinra should be used with caution in those with chronic kidney disease.

Anakinra is not specifically FDA approved for endometriosis. Although no data on its use in women with endometriosis have been published, there is no reason to expect women with endometriosis would be at any particular or increased risk than those in the general population.

This study is a randomized, double blinded, placebo controlled, cross-over clinical pilot study of 20 women. Patients diagnosed with surgical or imaging-technique proven endometriosis will be randomized to either treatment with an FDA approved medication (Anakinra) or a placebo. This is an investigator initiated single center study sponsored by the Swedish Orphan Biovitrum (SOBI). SOBI will provide the study drug and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 with regular menstrual periods every 24-32 days and not lasting more than 10 days per month
* Surgical or imaging proven endometriosis.
* At least a moderate level of menstrual pain based on the patient reported parameters of the B&B pain scale (>4/9) with dysmenorrhea being scored at least 2/3.
* Willing to remain on your current method of hormone therapy for duration of study

Exclusion Criteria:

* History of hysterectomy or oophorectomy.
* Non-response to GnRH agonist/antagonist, DMPA, aromatase inhibitors or danazol.
* Currently pregnant or attempting pregnancy.
* Contraindication to anakinra.
* Chronic kidney disease stage 4 and 5 or creatinine clearance <30mL/min/1.73m2.
* Abnormal LFTs, CBC or serum electrolytes including estimated GFR.
* Patient refusal.
* Plan to receive a live vaccine

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The primary aim of this study is to determine the impact of anakinra on menstrual pain due to endometriosis. Therefore, only women will be eligible for this study.
Enrollment: 20 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the impact of anakinra versus placebo on menstrual pain (dysmenorrhea) using the modified Biberoglu and Behrman scale. | Subjects will complete the baseline questionnaire at Visit 1. Subjects will fill out monthly questionnaires after the administration of either anakinra or placebo during 6 menstrual periods.
  The primary pain outcome measure is to determine the impact of anakinra on dysmenorrhea due to endometriosis, using the modified Biberoglu and Behrman scale. The modified Biberoglu and Behrman scale consists of three patient-reported symptoms (dysmenorrhea, dyspareunia, and non-menstrual pelvic pain). Each of these is separately graded on a scale from 0 to 3, with a max of 9 and higher numbers indicating more severe symptoms. Changes in dysmenorrhea is the primary endpoint.

SECONDARY OUTCOMES:
Comparison of the impact of anakinra versus placebo on dyspareunia and non menstrual pelvic pain using the modified Biberoglu and Behrman scale. | Subjects will complete the baseline questionnaire at Visit 1. Subjects will fill out monthly questionnaires after the administration of either anakinra or placebo during 6 menstrual periods.
  Secondary pain outcome measures are to determine the impact of anakinra on dyspareunia and non-menstrual pelvic pain due to endometriosis, using the modified Biberoglu and Behrman scale. The modified Biberoglu and Behrman scale consists of three patient-reported symptoms (dysmenorrhea, dyspareunia, and non-menstrual pelvic pain). Each of these is separately graded on a scale from 0 to 3, with a max of 9 and higher numbers indicating more severe symptoms. Changes in dyspareunia and non-menstrual pelvic pain are secondary pain endpoints.
Comparison of the impact of anakinra versus placebo on the quality of life using the Endometriosis Health Profile 30 questionnaire (EHP-30), conducted after each course of study medication administration. | Subjects will complete the baseline questionnaire at Visit 1. Subjects will fill out monthly questionnaires after the administration of either anakinra or placebo during 6 menstrual periods.
  The secondary outcome measure is to determine the impact of anakinra on the quality of life due to endometriosis, using the Endometriosis Health Profile 30 (EHP-30) questionnaire. The EHP-30 consists of a 30 item instrument that assesses pain, control and powerlessness, social support, emotional well-being, and self image. Each scale is standardized on a scale of 0 - 100, where 0 indicates the best health status through to 100 worst health status.
Comparison of serum inflammatory markers before and after anakinra administration. | There will be blood tests at the start and end of each of of the subject's next 6 menstrual periods for a total of 12 blood draws.
  The secondary outcome is to evaluate the effect of anakinra on serum inflammatory markers that are elevated in women with endometriosis. Relevant inflammatory markers of endometriosis include CRP, CA125, IL-1, IL-4, IL-6, IL-10, BDNF, Glycodelin, and ZAG. There will be blood tests at the start and end of each of of the subject's next 6 menstrual periods: At the time of each blood draw, we will collect 20 mL (approximately 4 teaspoons) of blood. This will be needed for each of the 6 study menstrual periods for a total of 12 blood draws. There will be a total of 240 ml of blood or approximately 16 tablespoons of blood collected throughout the entire study.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Agarwal, MD, Principal Investigator — UC San Diego
Locations (1):
- UCSD Reproductive Endocrinology, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
Only the PI, Dr. Foster and the study staff will have access to study subjects' research data.

REFERENCES:
- [Background] Kennedy S, Bergqvist A, Chapron C, D'Hooghe T, Dunselman G, Greb R, Hummelshoj L, Prentice A, Saridogan E; ESHRE Special Interest Group for Endometriosis and Endometrium Guideline Development Group. ESHRE guideline for the diagnosis and treatment of endometriosis. Hum Reprod. 2005 Oct;20(10):2698-704. doi: 10.1093/humrep/dei135. Epub 2005 Jun 24. PMID 15980014
- [Background] Khanaki K, Nouri M, Ardekani AM, Ghassemzadeh A, Shahnazi V, Sadeghi MR, Darabi M, Mehdizadeh A, Dolatkhah H, Saremi A, Imani AR, Rahimipour A. Evaluation of the relationship between endometriosis and omega-3 and omega-6 polyunsaturated fatty acids. Iran Biomed J. 2012;16(1):38-43. doi: 10.6091/ibj.1025.2012. PMID 22562031
- [Background] Marik JJ. Leuprolide acetate depot and hormonal add-back in endometriosis: a 12-month study. Obstet Gynecol. 1998 May;91(5 Pt 1):793-4. doi: 10.1097/00006250-199805000-00029. No abstract available. PMID 9572232
- [Background] Stratton P, Sinaii N, Segars J, Koziol D, Wesley R, Zimmer C, Winkel C, Nieman LK. Return of chronic pelvic pain from endometriosis after raloxifene treatment: a randomized controlled trial. Obstet Gynecol. 2008 Jan;111(1):88-96. doi: 10.1097/01.AOG.0000297307.35024.b5. PMID 18165396